CLINICAL TRIAL: NCT05920876
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Effectiveness of QLS32015 Injection in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of QLS32015 in Patients With Recurrent or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS32015-101
Record Dates: First submitted 2023-06-15; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS32015 (Experimental): Dose escalation and does expansion of QLS32015 injection will be evaluated.
  Interventions: Drug: QLS32015

INTERVENTIONS:
Drug: QLS32015 — Participants will receive subcutaneous (SC) injection of QLS32015. Eight dose groups were proposed, 21 days as a treatment cycle.
  Other Names: A Humanized GPRC5D x CD3 Bispecific Antibody

SUMMARY:
The purpose of this study is to characterize the safety of QLS32015 injection and to determine the recommended Phase 2 dose (RP2D) and to further evaluate the efficacy and safety of QLS32015 injection in participants with relapsed or refractory multiple myeloma at the recommended Phase 2 dose.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant disease with abnormal proliferation of clonal plasma cell, which is often accompanied by multiple osteolytic damage, hypercalcemia, anemia, and kidney damage. QLS32015 is a humanized immunoglobulin gamma-1 (IgG1) type bispecific antibody targeting G protein-coupled receptor family C group 5-member D (GPRC5D) and cluster of differentiation 3 (CD3). The study consists 3 periods: screening phase, treatment phase and a post-treatment follow-up phase. The study will evaluate safety, tolerability, pharmacokinetics and preliminary antitumor activity of QLS32015 administered to participants with relapsed or refractory multiple myeloma. Total duration of study is up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, regardless of gender.
* Subjects should be willing and able to comply with the study schedule and protocols.
* Documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria.
* Must have measurable disease as defined by the following: Serum M-protein greater than or equal to 1 g/dL; OR Urine M-protein greater than or equal to 200 mg/24 hours; OR Serum free light chain (FLC) assay; involved FLC level greater than or equal to 10 mg/dL provided the serum FLC ratio is abnormal.

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients of this product.
* Diagnosis of active plasma cell leukemia or systemic light chain amyloidosis.
* Has any active severe mental illness, medical illness, or other symptoms/conditions that may affect treatment, compliance, or the ability to provide informed consent, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Approximately 2 years
  Determination of the recommended phase 2 dose (RP2D) of QLS32015 injection in patient with relapsed or refractory multiple myeloma.
Incidence of adverse events（AEs） | Up to 2 years
  Assessing the incidence of adverse events (AEs) using the Common Terminology Criteria for Adverse Events (CTCAE Version 5).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years
  ORR assessed by the IMWG response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China